CLINICAL TRIAL: NCT02057289
Title: Micafungin Anti-Fungal Prophylaxis in Immunocompromised Pediatric Patients: A Pharmacokinetic Study
Brief Title: A Pharmacokinetic Study of Pediatric Micafungin Prophylaxis
Acronym: Micafungin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-4868
Record Dates: First submitted 2014-01-29; First posted 2014-02-07 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Immunocompromised; Bone Marrow Transplant; Cancer
Keywords: pediatric; antifungal; bone marrow; AML or relapsed ALL
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micafungin (Experimental): Subjects will be administered 5 mg/kg of micafungin intravenously as a ONE TIME dose.
  For patients undergoing Hematopoietic Stem Cell Transplant (HSCT), Micafungin will be given on during rest days (i.e. days when no chemotherapy is administered) and blood for pharmacokinetic measurements will be drawn over next 96 hours.
  Following this, further anti-fungal coverage will be at the discretion of the patient's attending physician. (I.e. other antifungal agent(s) or Micafungin at a standard clinical dose; repeat doses of 5mg/kg will NOT be administered.)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Micafungin (trade name Mycamine) is an echinocandin antifungal drug developed by Astellas Pharma. It inhibits the production of beta-1,3-glucan, an essential component of fungal cell walls. Micafungin is administered intravenously. It received final approval from the U.S. Food and Drug Administration on March 16, 2005, and gained approval in the European Union on April 25, 2008.
  Other Names: Mycamine

SUMMARY:
The purpose of this research study is to examine the pharmacokinetics (the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body) of micafungin when it is given at 5mg/kg dose to immunocompromised children as anti-fungal prophylaxis. These children are at high risk for developing invasive fungal disease due to their compromised immunity and associated variable degree and duration of neutropenia. Currently, children who receive micafungin are given daily or alternate day dosing. The investigators will give a ONE TIME dose of micafungin and draw PK levels up to 96 hours post-infusion. The investigators goal is to obtain comparable micafungin drug concentrations at the end of 96 hours (4 days) as compared to lower dose at every 24 hour dosing. The investigators dosing proposal is likely to be effective prophylaxis for immunocompromised patients and would broaden its applicability to larger populations.

DETAILED DESCRIPTION:
Disseminated fungal infection is a major cause of morbidity and mortality in immunocompromised children. Many of the drugs used for fungal prophylaxis have been associated with renal and hepatic toxicity. Also, breakthrough infections have been reported with the use of some of the oral agents due to poor oral absorption. An alternative approach is the use of intravenous micafungin for fungal prophylaxis. Micafungin has a distinct advantage due to its better safety profile, specifically in terms of hepatic and renal toxicity. Currently, children who receive micafungin are given daily or alternate day dosing (based on their last Pk study, Mehta et al 2010). The investigators objective is to examine the pharmacokinetics of micafungin when it is given on a less frequent schedule. The investigators hypothesize that a single dose of micafungin (at 5mg/kg) every 4 days will provide drug exposure equivalent to daily dosing (at 1mg/kg) while reducing administration costs and improving patient convenience (with essentially twice a week dosing regimen). Both animal and adult data support the use of this approach. Fifteen patients will be enrolled on this study and will be given a SINGLE DOSE of micafungin antifungal prophylaxis (5 mg/kg). Blood samples will be drawn for pharmacokinetic measurements after administration of micafungin. Plasma concentration data will be analyzed by compartmental and non-compartmental pharmacokinetic analysis. The data will also be analyzed by a population pharmacokinetic approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at risk for fungal infection and require prophylaxis. Example: patients undergoing blood and marrow transplant, immunodeficiency patients, patients with aplastic anemia.
* Age >= 6 months to <= 10 years (at time of enrollment).
* Patients with adequate organ function (documented within 2 weeks prior to start of micafungin):

  * Creatinine < 2 times upper limit normal
  * Total bilirubin and AST < 3 times upper limit normal

Exclusion Criteria:

* Patients who have history of past or evidence of active fungal disease (by either radiological studies or biopsy proven) or are being treated for presumed fungal infection.
* Patients who have history of allergy to micafungin or other echinocandin preparations, such as Caspofungin or Anidulafungin.
* Patients who have received micafungin or other echinocandin preparations in the previous two weeks.
* Patients receiving antifungal prophylaxis other than Fluconazole at the time of enrollment. This is due to the fact that during transplant, Fluconazole is usually switched to agents with better coverage. This will avoid the possibility of reducing effective antifungal coverage for the purpose of the study.
* Failure to sign informed consent, or inability to undergo informed consent process.
* It is not medically advisable to obtain the specimens necessary for this study.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics to measure the levels of micafungin | Prior to the micafungin infusion at hour 0, at the end of the infusion (60 min), then at 11/2, 2, 4, 6, 8, 10, 24, 36, 48, 60, 72, 84 and 96 hours after the start of the micafungin infusion.
  Blood samples from the above time points will be analyzed to study the bodily absorption, distribution, metabolism, and excretion of micafungin

CONTACTS AND LOCATIONS:
Overall Officials: Parinda Mehta, MD, Principal Investigator — CCHMC
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States